CLINICAL TRIAL: NCT00556777
Title: Phase 2 Study Evaluating the Feasibility and the Reproducibility of Concentrated Radiotherapy and Focalized Electrontherapy During Surgery for the Treatment of Older Patients With Breast Cancer
Brief Title: Radiation Therapy During Surgery in Treating Older Women With Stage I Breast Cancer
Acronym: IORT-Sein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000574074; CLCC-IORT-Sein; INCA-RECF0284
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Intervention Model Description: partial irradiation of the breast, after an enlarged tumorectomy and negative sentinel limph node, assessing the feasibility and technical reproducibility of a per-concentrated irradiationThe first treatment was a surgical operation focused on the initial tumor area as the only treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): breast conserving surgery with lymph node dissection + Intraoperative radiotherapy
  Interventions: Procedure: axillary lymph node dissection; Procedure: conventional surgery; Procedure: sentinel lymph node biopsy; Radiation: intraoperative radiation therapy

INTERVENTIONS:
Procedure: axillary lymph node dissection
Procedure: conventional surgery
Procedure: sentinel lymph node biopsy
Radiation: intraoperative radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Giving intraoperative radiation therapy may reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well giving radiation therapy during surgery works in treating older women with stage I breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Study the feasibility and reproducibility of intraoperative radiotherapy as the only treatment after lumpectomy in older women with stage I breast cancer.

Secondary

* Study the impact of this regimen on maintaining self-care.
* Study the quality of life (QLQ-C30) and satisfaction with care.
* Study regimen tolerance and cosmetic results.
* Evaluate the economic impact of this treatment.
* Study relapse-free and disease-specific survival.

OUTLINE: Patients undergo conservative breast surgery and axillary node dissection (sentinel node or classic resection). At this point, patients must have either negative axillary lymph nodes after removal of ≥ 6 lymph nodes, negative sentinel nodes, or have had a limited lumpectomy with negative margins ≥ 2 mm. Patients undergo intraoperative radiotherapy during surgery, before closing and reconstruction of the breast.

Patients may begin hormonal therapy after completing study therapy.

After completion of study therapy, patients are followed every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically confirmed stage I breast cancer

  * Size ≤ 20 mm (by ultrasound), N0, any quadrant
* Hormone receptor status not specified

Exclusion criteria:

* Distant metastases
* Inflammatory breast cancer
* Lobular in situ disease
* Invasive cancer or ductal carcinoma in situ
* Nonepithelial disease or sarcoma
* Multicentric disease
* Lymphatic embolism
* Margins of safety unknown or positive (in situ or invasive)
* Preoperative mammography showing diffuse microcalcification

PATIENT CHARACTERISTICS:

* Female
* Menopausal
* Karnofsky 70-100%
* No other prior cancer except basal cell skin cancer, uterine epithelioma in situ, or other cancer in complete remission for the past 5 years
* No geographic, social, or psychiatric reasons that would impede participation in study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior neoadjuvant therapy
* No concurrent participation in another study

Ages: 65 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-04-19 (Actual); Primary Completion 2008-12-31 (Actual); Study Completion 2008-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of feasibility of partial irradiation of the breast by per-operative electron therapy | During the treatment of irradiation (4 weeks)
  feasibility based on dosimetric criteria based on the Quality Index of the application.
Evaluation of reproducibility of partial irradiation of the breast by per-operative electron therapy | During the treatment of irradiation (4 weeks)
  reproducibility based on dosimetric criteria based on the Quality Index of the application.

SECONDARY OUTCOMES:
impact on Quality of life of partial irradiation of the breast by per-operative electron therapy | from the baseline to 12 months after the treatment
  Impact described by th scores of "Instrumental Activities of Daily Living scale"
impact on Quality of life of partial irradiation of the breast by per-operative electron therapy | from the baseline to 12 months after the treatment
  Impact described by th scores of "Activities of Daily Living scale"
Tolerability of partial irradiation of the breast by per-operative electron therapy | from the baseline to 12 months after the treatment
  Tolerability done with Common Terminology Criteria for Adverse Events scale
Relapse-free survival | from the baseline to 12 months after the treatment
  Relapse-free survival describes with radiologie evaluation
Disease-specific survival | from the baseline to 12 months after the treatment
  Relapse-free survival describes with radiologie evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Bernard Dubois, MD, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France

REFERENCES:
- [Background] Aaronson NK. Assessing the quality of life of patients in cancer clinical trials: Common problems and common sense solutions. Eur J Cancer. 1992;28A(8-9):1304-7. doi: 10.1016/0959-8049(92)90504-u. No abstract available. PMID 1515238
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Nattinger AB, Kneusel RT, Hoffmann RG, Gilligan MA. Relationship of distance from a radiotherapy facility and initial breast cancer treatment. J Natl Cancer Inst. 2001 Sep 5;93(17):1344-6. doi: 10.1093/jnci/93.17.1344. No abstract available. PMID 11535710
- [Background] Arnulf G. Lymphoedema of the upper limb after Halsted's operation of radical mastectomy.. Lymphography and phlebography. Therapeutic consequences. Vasc Surg. 1973 Jan-Feb;7(1):36-44. doi: 10.1177/153857447300700105. No abstract available. PMID 4691036
- [Background] Arriagada R, Le MG, Rochard F, Contesso G. Conservative treatment versus mastectomy in early breast cancer: patterns of failure with 15 years of follow-up data. Institut Gustave-Roussy Breast Cancer Group. J Clin Oncol. 1996 May;14(5):1558-64. doi: 10.1200/JCO.1996.14.5.1558. PMID 8622072
- [Background] Balducci L, Extermann M, Carreca I. Management of breast cancer in the older woman. Cancer Control. 2001 Sep-Oct;8(5):431-41. doi: 10.1177/107327480100800507. PMID 11579340
- [Background] Balducci L, Lyman GH. Cancer in the elderly. Epidemiologic and clinical implications. Clin Geriatr Med. 1997 Feb;13(1):1-14. PMID 8995097
- [Background] Ballard-Barbash R, Potosky AL, Harlan LC, Nayfield SG, Kessler LG. Factors associated with surgical and radiation therapy for early stage breast cancer in older women. J Natl Cancer Inst. 1996 Jun 5;88(11):716-26. doi: 10.1093/jnci/88.11.716. PMID 8637025
- [Background] Bartelink H, Horiot JC, Poortmans P, Struikmans H, Van den Bogaert W, Barillot I, Fourquet A, Borger J, Jager J, Hoogenraad W, Collette L, Pierart M; European Organization for Research and Treatment of Cancer Radiotherapy and Breast Cancer Groups. Recurrence rates after treatment of breast cancer with standard radiotherapy with or without additional radiation. N Engl J Med. 2001 Nov 8;345(19):1378-87. doi: 10.1056/NEJMoa010874. PMID 11794170
- [Background] Bates T, Riley DL, Houghton J, Fallowfield L, Baum M. Breast cancer in elderly women: a Cancer Research Campaign trial comparing treatment with tamoxifen and optimal surgery with tamoxifen alone. The Elderly Breast Cancer Working Party. Br J Surg. 1991 May;78(5):591-4. doi: 10.1002/bjs.1800780523. PMID 2059815
- [Background] Brenier JL. The role of the Halsted operation in treatment of breast cancer. Int Surg. 1967 Mar;47(3):288-90. No abstract available. PMID 4962239
- [Background] Buchholz TA, Austin-Seymour MM, Moe RE, Ellis GK, Livingston RB, Pelton JG, Griffin TW. Effect of delay in radiation in the combined modality treatment of breast cancer. Int J Radiat Oncol Biol Phys. 1993 Apr 30;26(1):23-35. doi: 10.1016/0360-3016(93)90169-v. PMID 8482628
- [Background] Clark RM, Whelan T, Levine M, Roberts R, Willan A, McCulloch P, Lipa M, Wilkinson RH, Mahoney LJ. Randomized clinical trial of breast irradiation following lumpectomy and axillary dissection for node-negative breast cancer: an update. Ontario Clinical Oncology Group. J Natl Cancer Inst. 1996 Nov 20;88(22):1659-64. doi: 10.1093/jnci/88.22.1659. PMID 8931610
- [Background] Cooke AL, Perera F, Fisher B, Opeitum A, Yu N. Tamoxifen with and without radiation after partial mastectomy in patients with involved nodes. Int J Radiat Oncol Biol Phys. 1995 Feb 15;31(4):777-81. doi: 10.1016/0360-3016(94)00499-4. PMID 7860388
- [Background] Diab SG, Elledge RM, Clark GM. Tumor characteristics and clinical outcome of elderly women with breast cancer. J Natl Cancer Inst. 2000 Apr 5;92(7):550-6. doi: 10.1093/jnci/92.7.550. PMID 10749910
- [Background] Dinh QC. [The population of France up to 2050]. Econ Stat. 1994;(274):7-32, 93, 95,. French. PMID 12346113
- [Background] Fentiman IS, Poole C, Tong D, Winter PJ, Gregory WM, Mayles HM, Turner P, Chaudary MA, Rubens RD. Inadequacy of iridium implant as sole radiation treatment for operable breast cancer. Eur J Cancer. 1996 Apr;32A(4):608-11. doi: 10.1016/0959-8049(95)00639-7. PMID 8695261
- [Background] Fentiman IS, Poole C, Tong D, Winter PJ, Mayles HM, Turner P, Chaudary MA, Rubens RD. Iridium implant treatment without external radiotherapy for operable breast cancer: a pilot study. Eur J Cancer. 1991;27(4):447-50. doi: 10.1016/0277-5379(91)90383-o. PMID 1827719
- [Background] Fisher B, Anderson S, Redmond CK, Wolmark N, Wickerham DL, Cronin WM. Reanalysis and results after 12 years of follow-up in a randomized clinical trial comparing total mastectomy with lumpectomy with or without irradiation in the treatment of breast cancer. N Engl J Med. 1995 Nov 30;333(22):1456-61. doi: 10.1056/NEJM199511303332203. PMID 7477145
- [Background] Fisher B, Anderson S. Conservative surgery for the management of invasive and noninvasive carcinoma of the breast: NSABP trials. National Surgical Adjuvant Breast and Bowel Project. World J Surg. 1994 Jan-Feb;18(1):63-9. doi: 10.1007/BF00348193. PMID 8197778
- [Background] Fisher B, Costantino J, Redmond C, Fisher E, Margolese R, Dimitrov N, Wolmark N, Wickerham DL, Deutsch M, Ore L, et al. Lumpectomy compared with lumpectomy and radiation therapy for the treatment of intraductal breast cancer. N Engl J Med. 1993 Jun 3;328(22):1581-6. doi: 10.1056/NEJM199306033282201. PMID 8292119
- [Background] Fisher B, Redmond C, Poisson R, Margolese R, Wolmark N, Wickerham L, Fisher E, Deutsch M, Caplan R, Pilch Y, et al. Eight-year results of a randomized clinical trial comparing total mastectomy and lumpectomy with or without irradiation in the treatment of breast cancer. N Engl J Med. 1989 Mar 30;320(13):822-8. doi: 10.1056/NEJM198903303201302. PMID 2927449
- [Background] Forrest AP, Stewart HJ, Everington D, Prescott RJ, McArdle CS, Harnett AN, Smith DC, George WD. Randomised controlled trial of conservation therapy for breast cancer: 6-year analysis of the Scottish trial. Scottish Cancer Trials Breast Group. Lancet. 1996 Sep 14;348(9029):708-13. doi: 10.1016/s0140-6736(96)02133-2. PMID 8806289
- [Background] Fowble B. An assessment of treatment options for breast conservation in the elderly woman with early stage breast cancer. Int J Radiat Oncol Biol Phys. 1995 Feb 15;31(4):1015-7. doi: 10.1016/0360-3016(95)00008-9. No abstract available. PMID 7860374
- [Background] Gazet JC, Ford HT, Coombes RC, Bland JM, Sutcliffe R, Quilliam J, Lowndes S. Prospective randomized trial of tamoxifen vs surgery in elderly patients with breast cancer. Eur J Surg Oncol. 1994 Jun;20(3):207-14. PMID 8181594
- [Background] Gruenberger T, Gorlitzer M, Soliman T, Rudas M, Mittlboeck M, Gnant M, Reiner A, Teleky B, Seitz W, Jakesz R. It is possible to omit postoperative irradiation in a highly selected group of elderly breast cancer patients. Breast Cancer Res Treat. 1998 Jul;50(1):37-46. doi: 10.1023/a:1006064608360. PMID 9802618
- [Background] Harms W, Krempien R, Hensley FW, Berns C, Wannenmacher M, Fritz P. Results of chest wall reirradiation using pulsed-dose-rate (PDR) brachytherapy molds for breast cancer local recurrences. Int J Radiat Oncol Biol Phys. 2001 Jan 1;49(1):205-10. doi: 10.1016/s0360-3016(00)01360-2. PMID 11163516
- [Background] Hebert-Croteau N, Brisson J, Latreille J, Blanchette C, Deschenes L. Compliance with consensus recommendations for the treatment of early stage breast carcinoma in elderly women. Cancer. 1999 Mar 1;85(5):1104-13. PMID 10091795
- [Background] Holland R, Connolly JL, Gelman R, Mravunac M, Hendriks JH, Verbeek AL, Schnitt SJ, Silver B, Boyages J, Harris JR. The presence of an extensive intraductal component following a limited excision correlates with prominent residual disease in the remainder of the breast. J Clin Oncol. 1990 Jan;8(1):113-8. doi: 10.1200/JCO.1990.8.1.113. PMID 2153190
- [Background] Holland R, Veling SH, Mravunac M, Hendriks JH. Histologic multifocality of Tis, T1-2 breast carcinomas. Implications for clinical trials of breast-conserving surgery. Cancer. 1985 Sep 1;56(5):979-90. doi: 10.1002/1097-0142(19850901)56:53.0.co;2-n. PMID 2990668
- [Background] Jacobson JA, Danforth DN, Cowan KH, d'Angelo T, Steinberg SM, Pierce L, Lippman ME, Lichter AS, Glatstein E, Okunieff P. Ten-year results of a comparison of conservation with mastectomy in the treatment of stage I and II breast cancer. N Engl J Med. 1995 Apr 6;332(14):907-11. doi: 10.1056/NEJM199504063321402. PMID 7877647
- [Background] Kantorowitz DA, Poulter CA, Sischy B, Paterson E, Sobel SH, Rubin P, Dvoretsky PA, Mishalak W, Doane KL. Treatment of breast cancer among elderly women with segmental mastectomy or segmental mastectomy plus postoperative radiotherapy. Int J Radiat Oncol Biol Phys. 1988 Aug;15(2):263-70. doi: 10.1016/s0360-3016(98)90003-7. PMID 3403309
- [Background] Katz S, Downs TD, Cash HR, Grotz RC. Progress in development of the index of ADL. Gerontologist. 1970 Spring;10(1):20-30. doi: 10.1093/geront/10.1_part_1.20. No abstract available. PMID 5420677
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Background] King TA, Bolton JS, Kuske RR, Fuhrman GM, Scroggins TG, Jiang XZ. Long-term results of wide-field brachytherapy as the sole method of radiation therapy after segmental mastectomy for T(is,1,2) breast cancer. Am J Surg. 2000 Oct;180(4):299-304. doi: 10.1016/s0002-9610(00)00454-2. PMID 11113440
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Leonard CE, Wood ME, Zhen B, Rankin J, Waitz DA, Norton L, Howell K, Sedlacek S. Does administration of chemotherapy before radiotherapy in breast cancer patients treated with conservative surgery negatively impact local control? J Clin Oncol. 1995 Dec;13(12):2906-15. doi: 10.1200/JCO.1995.13.12.2906. PMID 8523054
- [Background] Liljegren G, Holmberg L, Bergh J, Lindgren A, Tabar L, Nordgren H, Adami HO. 10-Year results after sector resection with or without postoperative radiotherapy for stage I breast cancer: a randomized trial. J Clin Oncol. 1999 Aug;17(8):2326-33. doi: 10.1200/JCO.1999.17.8.2326. PMID 10561294
- [Background] Maddox WA, Carpenter JT Jr, Laws HL, Soong SJ, Cloud G, Urist MM, Balch CM. A randomized prospective trial of radical (Halsted) mastectomy versus modified radical mastectomy in 311 breast cancer patients. Ann Surg. 1983 Aug;198(2):207-12. doi: 10.1097/00000658-198308000-00016. PMID 6870379
- [Background] Macquart-Moulin G, Viens P, Bouscary ML, Genre D, Resbeut M, Gravis G, Camerlo J, Maraninchi D, Moatti JP. Discordance between physicians' estimations and breast cancer patients' self-assessment of side-effects of chemotherapy: an issue for quality of care. Br J Cancer. 1997;76(12):1640-5. doi: 10.1038/bjc.1997.610. PMID 9413955
- [Background] Macquart-Moulin G, Viens P, Genre D, Bouscary ML, Resbeut M, Gravis G, Camerlo J, Maraninchi D, Moatti JP. Concomitant chemoradiotherapy for patients with nonmetastatic breast carcinoma: side effects, quality of life, and organization. Cancer. 1999 May 15;85(10):2190-9. PMID 10326697
- [Background] Mandelblatt JS, Hadley J, Kerner JF, Schulman KA, Gold K, Dunmore-Griffith J, Edge S, Guadagnoli E, Lynch JJ, Meropol NJ, Weeks JC, Winn R. Patterns of breast carcinoma treatment in older women: patient preference and clinical and physical influences. Cancer. 2000 Aug 1;89(3):561-73. PMID 10931455
- [Background] Morimoto T, Okazaki K, Komaki K, Sasa M, Mori T, Tsuzuki H, Kamamura Y, Miki H, Monden Y. Cancerous residue in breast-conserving surgery. J Surg Oncol. 1993 Feb;52(2):71-6. doi: 10.1002/jso.2930520203. PMID 8385722
- [Background] Nemoto T, Dao TL. Is modified radical mastectomy adequate for axillary lymph node dissection? Ann Surg. 1975 Dec;182(6):722-3. doi: 10.1097/00000658-197512000-00011. PMID 1190875
- [Background] Nemoto T, Patel JK, Rosner D, Dao TL, Schuh M, Penetrante R. Factors affecting recurrence in lumpectomy without irradiation for breast cancer. Cancer. 1991 Apr 15;67(8):2079-82. doi: 10.1002/1097-0142(19910415)67:83.0.co;2-s. PMID 1848474
- [Background] Favourable and unfavourable effects on long-term survival of radiotherapy for early breast cancer: an overview of the randomised trials. Early Breast Cancer Trialists' Collaborative Group. Lancet. 2000 May 20;355(9217):1757-70. PMID 10832826
- [Background] Perera F, Engel J, Holliday R, Scott L, Girotti M, Girvan D, Chisela F, Venkatesan V. Local resection and brachytherapy confined to the lumpectomy site for early breast cancer: a pilot study. J Surg Oncol. 1997 Aug;65(4):263-7; discussion 267-8. doi: 10.1002/(sici)1096-9098(199708)65:43.0.co;2-3. PMID 9274791
- [Background] Ravitch MM. Carcinoma of the breast: the place of the Halsted radical mastectomy. Johns Hopkins Med J. 1971 Oct;129(4):202-11. No abstract available. PMID 4950576
- [Background] Reed MW, Morrison JM. Wide local excision as the sole primary treatment in elderly patients with carcinoma of the breast. Br J Surg. 1989 Sep;76(9):898-900. doi: 10.1002/bjs.1800760908. PMID 2804582
- [Background] Romestaing P, Lehingue Y, Carrie C, Coquard R, Montbarbon X, Ardiet JM, Mamelle N, Gerard JP. Role of a 10-Gy boost in the conservative treatment of early breast cancer: results of a randomized clinical trial in Lyon, France. J Clin Oncol. 1997 Mar;15(3):963-8. doi: 10.1200/JCO.1997.15.3.963. PMID 9060534
- [Background] Silliman RA, Balducci L, Goodwin JS, Holmes FF, Leventhal EA. Breast cancer care in old age: what we know, don't know, and do. J Natl Cancer Inst. 1993 Feb 3;85(3):190-9. doi: 10.1093/jnci/85.3.190. PMID 8423623
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Sminia P, Schneider CJ, van Tienhoven G, Koedooder K, Blank LE, Gonzalez Gonzalez D. Office hours pulsed brachytherapy boost in breast cancer. Radiother Oncol. 2001 Jun;59(3):273-80. doi: 10.1016/s0167-8140(01)00335-8. PMID 11369068
- [Background] Smith TE, Lee D, Turner BC, Carter D, Haffty BG. True recurrence vs. new primary ipsilateral breast tumor relapse: an analysis of clinical and pathologic differences and their implications in natural history, prognoses, and therapeutic management. Int J Radiat Oncol Biol Phys. 2000 Dec 1;48(5):1281-9. doi: 10.1016/s0360-3016(00)01378-x. PMID 11121624
- [Background] Solin LJ, Schultz DJ, Fowble BL. Ten-year results of the treatment of early-stage breast carcinoma in elderly women using breast-conserving surgery and definitive breast irradiation. Int J Radiat Oncol Biol Phys. 1995 Aug 30;33(1):45-51. doi: 10.1016/0360-3016(95)00104-7. PMID 7642430
- [Background] Sprangers MA, Groenvold M, Arraras JI, Franklin J, te Velde A, Muller M, Franzini L, Williams A, de Haes HC, Hopwood P, Cull A, Aaronson NK. The European Organization for Research and Treatment of Cancer breast cancer-specific quality-of-life questionnaire module: first results from a three-country field study. J Clin Oncol. 1996 Oct;14(10):2756-68. doi: 10.1200/JCO.1996.14.10.2756. PMID 8874337
- [Background] Vaidya JS, Baum M, Tobias JS, D'Souza DP, Naidu SV, Morgan S, Metaxas M, Harte KJ, Sliski AP, Thomson E. Targeted intra-operative radiotherapy (Targit): an innovative method of treatment for early breast cancer. Ann Oncol. 2001 Aug;12(8):1075-80. doi: 10.1023/a:1011609401132. PMID 11583188
- [Background] van Dongen JA, Voogd AC, Fentiman IS, Legrand C, Sylvester RJ, Tong D, van der Schueren E, Helle PA, van Zijl K, Bartelink H. Long-term results of a randomized trial comparing breast-conserving therapy with mastectomy: European Organization for Research and Treatment of Cancer 10801 trial. J Natl Cancer Inst. 2000 Jul 19;92(14):1143-50. doi: 10.1093/jnci/92.14.1143. PMID 10904087
- [Background] Veronesi U, Saccozzi R, Del Vecchio M, Banfi A, Clemente C, De Lena M, Gallus G, Greco M, Luini A, Marubini E, Muscolino G, Rilke F, Salvadori B, Zecchini A, Zucali R. Comparing radical mastectomy with quadrantectomy, axillary dissection, and radiotherapy in patients with small cancers of the breast. N Engl J Med. 1981 Jul 2;305(1):6-11. doi: 10.1056/NEJM198107023050102. PMID 7015141
- [Background] Veronesi U, Luini A, Del Vecchio M, Greco M, Galimberti V, Merson M, Rilke F, Sacchini V, Saccozzi R, Savio T, et al. Radiotherapy after breast-preserving surgery in women with localized cancer of the breast. N Engl J Med. 1993 Jun 3;328(22):1587-91. doi: 10.1056/NEJM199306033282202. PMID 8387637
- [Background] Veronesi U, Marubini E, Mariani L, Galimberti V, Luini A, Veronesi P, Salvadori B, Zucali R. Radiotherapy after breast-conserving surgery in small breast carcinoma: long-term results of a randomized trial. Ann Oncol. 2001 Jul;12(7):997-1003. doi: 10.1023/a:1011136326943. PMID 11521809
- [Background] Vicini F, Kini VR, Chen P, Horwitz E, Gustafson G, Benitez P, Edmundson G, Goldstein N, McCarthy K, Martinez A. Irradiation of the tumor bed alone after lumpectomy in selected patients with early-stage breast cancer treated with breast conserving therapy. J Surg Oncol. 1999 Jan;70(1):33-40. doi: 10.1002/(sici)1096-9098(199901)70:13.0.co;2-o. PMID 9989418
- [Background] Vicini FA, Baglan KL, Kestin LL, Mitchell C, Chen PY, Frazier RC, Edmundson G, Goldstein NS, Benitez P, Huang RR, Martinez A. Accelerated treatment of breast cancer. J Clin Oncol. 2001 Apr 1;19(7):1993-2001. doi: 10.1200/JCO.2001.19.7.1993. PMID 11283132
- [Background] Vicini FA, Kestin LL, Goldstein NS, Baglan KL, Pettinga JE, Martinez AA. Relationship between excision volume, margin status, and tumor size with the development of local recurrence in patients with ductal carcinoma-in-situ treated with breast-conserving therapy. J Surg Oncol. 2001 Apr;76(4):245-54. doi: 10.1002/jso.1041. PMID 11320515
- [Background] Vlastos G, Mirza NQ, Meric F, Hunt KK, Kuerer HM, Ames FC, Ross MI, Buchholz TA, Hortobagyi GN, Singletary SE. Breast conservation therapy as a treatment option for the elderly. The M. D. Anderson experience. Cancer. 2001 Sep 1;92(5):1092-100. doi: 10.1002/1097-0142(20010901)92:53.0.co;2-p. PMID 11571720
- [Background] von Rueden DG, Sessions SC. Alternative therapy for elderly patients with breast cancer. Am Surg. 1994 Jan;60(1):72-8. PMID 8273979
- [Background] William Stewart Halsted (1852-1922) surgeon of the "Hopkins Four". JAMA. 1970 Sep 21;213(12):2072-4. No abstract available. PMID 4916652